CLINICAL TRIAL: NCT04825795
Title: Effect of DPP4 Inhibitors on Coronary Atherosclerosis in Patients With Diabetes Mellitus on Insulin Therapy
Brief Title: DPP4 Inhibitor and Coronary Atherosclerosis in Patients Receiving Insulin Therapy
Status: Completed | Type: Observational
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Sang Hyun Ihm, MD PhD, Professor, The Catholic University of Korea
Other Study IDs: XC21WIDI0044
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Dipeptidyl-Peptidase IV Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DPP4-inhibitor: Patients who were prescribed DPP4-inhibitor during the period between two coronary CT scan.
  Interventions: Drug: DPP4-inhibitor
- No DPP4-inhibitor: Patients who were not prescribed DPP4-inhibitor during the period between two coronary CT scan.
  Interventions: Drug: No DPP4-inhibitor

INTERVENTIONS:
Drug: DPP4-inhibitor — Prescription of DPP4-inhibitor during the period between the two coronary CT scan
  Groups: DPP4-inhibitor
Drug: No DPP4-inhibitor — No prescription of DPP4-inhibitor during the period between the two coronary CT scan
  Groups: No DPP4-inhibitor

SUMMARY:
The study aim is to evaluate whether DPP4-inhibitor could reduce coronary atherosclerosis assessed by CT scan in patients receiving insulin for diabetes mellitus. In this retrospective study, changes in obstructive coronary artery disease prevalence and coronary calcium burden between two coronary CT scans will be compared in patients with and without receiving DPP4-inhibitor.

DETAILED DESCRIPTION:
This is a retrospective study using medical records in two hospitals affiliated to the Catholic University of Korea. Patients with diabetes mellitus who received insulin are retrospectively enrolled. Among those, only patients who underwent coronary CT scan for more than two times will be included. Included patients will be classified into DPP4-inhibitor group and no DPP4-inhibitor group according to the prescribed medication. The changes in obstructive coronary artery disease prevalence and coronary calcium score per one year will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus
* Receiving chronic insulin therapy (prescription of insulin pen)
* Who underwent more than 2 times of coronary CT scan

Exclusion Criteria:

* Age <18

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were diagnosed with diabetes mellitus and receiving chronic insulin therapy will be enrolled. Among those, only patients who underwent more than two times of coronary CT scan will be included.
Sampling Method: Non-Probability Sample
Enrollment: 4007 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of obstructive coronary disease | one year
  Change in the prevalence of obstructive coronary disease, defined as >50 percent stenosis in coronary CT scan

SECONDARY OUTCOMES:
Change in coronary calcium score | one year
  Change in coronary calcium score, measured by two coronary CT scan per one year.
  Agatston score has minumum value of 0 and no maximum vavlue. Higher agatston score indicated severe calcification and worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Hyun Ihm, MD,PhD, Principal Investigator — Bucheon St. Mary's Hospital, College of Medicine, The Catholic University of Korea
Locations (1):
- Bucheon St. Mary's Hospital, Bucheon-si, South Korea

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data, because the clinical medical records using in this study are not open to public.